CLINICAL TRIAL: NCT01162096
Title: A Two Step Approach To Non-Myeloablative Matched-Sibling Allogeneic Hematopoietic Stem Cell Transplantation for Hematological Malignancies
Brief Title: Reduced Intensity Haploidentical Transplant for Hematological Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06U.328; 2006-29 (Other: CCRRC); JT 1149 (Other: JeffTrial Number)
Record Dates: First submitted 2010-07-12; First posted 2010-07-14 (Estimated); Results first posted 2015-01-15 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Hematological Malignancies
Keywords: Reduced Intensity Haploidentical Transplant
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transplantation (Experimental)
  Interventions: Device: Haploidentical Allogeneic Transplantation

INTERVENTIONS:
Device: Haploidentical Allogeneic Transplantation — Patients undergoing reduced intensity haploidentical hematopoietic stem cell transplant from a partially matched related donor.
  Other Names: CliniMACS

SUMMARY:
Many patients with hematological malignancies (leukemia, lymphoma, multiple myeloma) cannot undergo hematopoietic stem cell transplantation (HSCT) because they do not have a well matched donor. HSCT from partially matched family donors (haploidentical HSCT) is an option for most patients but has been associated with poor outcomes. This study was designed to test whether using an exact amount of a donor's lymphocytes (white cells) and dividing the transplant process into 2 steps, would increase overall survival by decreasing complications. The therapy is reduced intensity so it is targeted, but not limited to, patients over the age of 65 or those who have had previous transplants.

DETAILED DESCRIPTION:
Haploidentical hematopoietic stem cell transplant is a life saving therapy for patients who are without well matched donors. This type of therapy has been associated with poor outcomes in the past due to complications such as infection. The Jefferson 2 Step approach was designed to allow the infusion of an exact dose of tolerized lymphocytes in haploidentical transplant in order to allow for immune reconstitution post transplant to avoid infectious complications while still having acceptable rates of GVHD. In this approach, older patients or patients who were transplanted previously with high-risk hematological malignancies undergo chemotherapy with fludarabine and cytarabine or thiotepa. The patients then receive an exact dose of their donors' lymphocytes. The phase I portion of the study determined the optimal dose of lymphocytes. Two days after receiving the donor lymphocytes, the patients receive 2 daily doses of cyclophosphamide. The purpose of the cyclophosphamide is for in-vivo tolerization of the lymphocytes. One day after receiving cyclophosphamide, the patients receive stem cell from their donor. Tacrolimus and mycophenolate mofetil are used as GVHD prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient with a hematologic or oncologic diagnosis in which allogeneic HSCT is thought to be beneficial, and in whom front-line therapy has already been applied.
2. Patients must have a related donor who is a two or more allele mismatch at the HLA-A;B; C; DR loci.
3. Patients who have sibling donors with a one antigen mismatch due to recombination will not be enrolled in this protocol.
4. Patients must adequate organ function:

   1. LVEF of >45%
   2. DLCO >45% of predicted corrected for hemoglobin
   3. Adequate liver function as defined by a serum bilirubin <1.8, AST or ALT < 2.5X upper limit of normal
   4. Serum creatinine < 2.0 mg/dl or creatinine clearance of > 40 ml/min
5. Performance status > 70% (Karnofsky)
6. Patients must be willing to use contraception if they have childbearing potential
7. Able to give informed consent

Exclusion Criteria:

1. Performance status of < 70% (Karnofsky)
2. HIV positive
3. Active involvement of the central nervous system with malignancy
4. Psychiatric disorder that would preclude patients from signing an informed consent
5. Pregnancy
6. Patients with life expectancy of < 6 months for reasons other than their underlying hematologic/oncologic disorder or complications there from.
7. Patients who have received alemtuzumab within 8 weeks of transplant admission, or who have recently received horse or rabbit anti-thymocyte globulin and have ATG levels of > 2 µgm/ml.
8. Patients who cannot receive cyclophosphamide
9. Patients with evidence of another malignancy, exclusive of a skin cancer that requires only local treatment, should not be enrolled on this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-09; Primary Completion 2010-09 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Flomenberg, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transplantation
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Transplantation
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.23 (15.57)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival at 6 Months Post-transplant in Patients Receiving a Partially-matched Related Donor Allogeneic Transplant After Reduced-intensity Conditioning
Description: Number of patients alive at 6 months post-transplant
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Transplantation
Number analyzed (Participants) | 34
Participants | 22

2. Secondary Outcome: Number of Participants With Successful Engraftment
Time Frame: 6 months
Population: 32 patients are evaluable for engraftment
Measure: Count of Participants; unit: Participants
Arm/Group | Transplantation
Number analyzed (Participants) | 32
Participants | 31

3. Secondary Outcome: Immune Reconstitution
Time Frame: Up to 5 years
Measure: Median (Full Range); unit: cells/ul
Arm/Group | Transplantation
Number analyzed (Participants) | 34
cells/ul
  CD3/4 count at day 28 | 35.945 [2.1 to 213.6]
  CD3/4 count at day 90 | 104.540 [22.4 to 424.2]
  CD3/8 count at day 28 | 26.50 [2.1 to 213.6]
  CD3/8 count at day 90 | 119.2 [11.2 to 849.6]

ADVERSE EVENTS:
Arm/Group | Transplantation
Serious Adverse Events (participants affected / at risk) | 14/34
Other Adverse Events (participants affected / at risk) | 0/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transplantation (N=34)
Death - Multi-organ failure (General disorders) | 3 (3)
Death - Disease progression NOS (General disorders) | 6 (6)
Death - Death NOS (General disorders) | 5 (5)
Opportunistic infection associated with >=Grade 2 Lymphopenia (Infections and infestations) | 9 (12)
Infection - Other (Infections and infestations) | 5 (5)
Blood/Bone Marrow - other (Blood and lymphatic system disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Cardiac General - other (Cardiac disorders) | 2 (2)
Hypotension (Cardiac disorders) | 3 (3)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Allergic reaction/ hypersensitivity (Immune system disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1)
Left ventricular diastolic dysfunction (Cardiac disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastrointestinal - other (Gastrointestinal disorders) | 1 (1)
Myelitis (Nervous system disorders) | 1 (1)
Pulmonary/Upper Respiratory - other (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes